CLINICAL TRIAL: NCT05136443
Title: Prospective Analysis of Loteprednol Etabonate Ophthalmic Suspension 0.25% for Prevention of Immunologic Rejection After Descemet Membrane Endothelial Keratoplasty
Brief Title: Loteprednol Etabonate 0.25% for Prevention of Cornea Transplant Rejection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Price Vision Group (Industry)
Collaborators: Kala Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-002
Record Dates: First submitted 2021-10-29; First posted 2021-11-29 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2023-09

CONDITIONS: Corneal Endothelial Dystrophy; Corneal Edema
MeSH Terms: conditions — Corneal Dystrophy, Posterior Polymorphous, 1; Corneal Edema | interventions — Loteprednol Etabonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Preventative Treatment (Experimental): Loteprednol etabonate ophthalmic suspension 0.25% dosed 4 times daily for 2 months, 3 times daily for one month, twice daily for one month, and once daily until the 1 year postop exam.
  Interventions: Drug: loteprednol etabonate 0.25% ophthalmic suspension

INTERVENTIONS:
Drug: loteprednol etabonate 0.25% ophthalmic suspension — tapering dose
  Other Names: Eysuvis

SUMMARY:
The purpose of this study is to assess off-label use of loteprednol etabonate 0.25% ophthalmic suspension (Eysuvis) for prevention of immunologic rejection in the first year after Descemet membrane endothelial keratoplasty (DMEK). Topical corticosteroids have long been the mainstay for preventing and treating cornea transplant rejection although none are specifically approved for this purpose. The rates of immunologic rejection episodes and steroid-induced ocular hypertension will be compared with the respective rates observed in earlier studies with prednisolone acetate 1% suspension, loteprednol etabonate 0.5% gel, and fluorometholone 0.1% suspension after DMEK.

ELIGIBILITY:
Inclusion Criteria:

* o At least 18 years of age

  * Male or female patient who had DMEK within the past 1 to 7 weeks.
  * Patient is able and willing to administer eye drops.
  * Patient is able to comprehend and has signed the Informed Consent form.
  * Patient is likely to complete the 11-month study duration.

Exclusion Criteria:

* o A history of a previous rejection episode in the study eye

  * A patient exhibiting intraocular inflammation.
  * A patient with a known sensitivity to any of the ingredients in the study medications
  * A patient who has a condition (i.e., UNCONTROLLED systemic disease) or is in a situation which in the investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study
  * A patient with abnormal eyelid function.
  * A patient that is exhibiting active corneal ulceration, keratitis, or conjunctivitis, or who has a history of herpetic keratitis.
  * Presence of any ocular disease that would interfere with the evaluation of the study treatment. However, patients with a history of cystoid macular edema, age-related macular degeneration, controlled glaucoma, corneal neovascularization, and other non-interfering comorbidities may be enrolled.
  * A patient with a history of non-compliance with using prescribed medication.
  * Patients who are pregnant or planning to become pregnant within the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, Jr., MD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Price MO, Feng MT, Scanameo A, Price FW Jr. Loteprednol Etabonate 0.5% Gel Vs. Prednisolone Acetate 1% Solution After Descemet Membrane Endothelial Keratoplasty: Prospective Randomized Trial. Cornea. 2015 Aug;34(8):853-8. doi: 10.1097/ICO.0000000000000475. PMID 26020827
- [Background] Price MO, Price FW Jr, Kruse FE, Bachmann BO, Tourtas T. Randomized comparison of topical prednisolone acetate 1% versus fluorometholone 0.1% in the first year after descemet membrane endothelial keratoplasty. Cornea. 2014 Sep;33(9):880-6. doi: 10.1097/ICO.0000000000000206. PMID 25062336
- [Result] Price MO, Feng MT, Gang A, Price FW Jr. Prospective Assessment of Loteprednol Etabonate 0.25% for Prevention of Immunologic Rejection After Descemet Membrane Endothelial Keratoplasty in Eyes With Fuchs Dystrophy. Cornea. 2024 Aug 1;43(8):1028-1030. doi: 10.1097/ICO.0000000000003398. Epub 2023 Sep 21. PMID 37733966

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preventative Treatment
Started | 70
Completed | 66
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Preventative Treatment
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 70 [29 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Immunologic Rejection
Description: incidence of immunologic rejection episodes
Time Frame: 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | Preventative Treatment
Number analyzed (Participants) | 70
Participants | 0

2. Primary Outcome: Steroid-induced Ocular Hypertension
Description: incidence of steroid-induced ocular hypertension
Time Frame: 11 months
Measure: Count of Participants; unit: Participants
Arm/Group | Preventative Treatment
Number analyzed (Participants) | 70
Participants | 1

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Preventative Treatment
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 3/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preventative Treatment (N=70)
Steroid induced intraocular pressure elevation (Eye disorders) | 1 (1)
Instillation site discomfort (Eye disorders) | 2 (2) — Ocular discomfort associated with instillation of study eye drop

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT05136443/Prot_SAP_000.pdf